CLINICAL TRIAL: NCT05970224
Title: A Phase IIa, Randomized, Open-label, Proof-of-Concept Study to Evaluate Safety, Tolerability and Efficacy of Ir-CPI in Patients With Spontaneous Intracerebral Haemorrhage
Brief Title: A Study to Evaluate the Safety, Tolerability and the Effects of Ixodes Ricinus-Contact Phase Inhibitor (Ir-CPI) in Adult Patients With Spontaneous Intracerebral Haemorrhage
Acronym: BIRCH
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Bioxodes S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Clin_IrCPI_201; 2022-500491-53-00 (Registry Identifier: CTIS)
Record Dates: First submitted 2023-07-24; First posted 2023-08-01 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-04

CONDITIONS: Intracerebral Hemorrhage
Keywords: Ir-CPI; ICH; Secondary brain injury; Ixodes ricinus-Contact Phase Inhibitor; Neutrophil; Antithrombotic; Intracranial hemorrhage; Stroke; Brain; Inflammation; Neuroinflammation; Cerebrovascular disorders
MeSH Terms: conditions — Cerebral Hemorrhage; Intracranial Hemorrhages; Stroke; Inflammation; Neuroinflammatory Diseases; Cerebrovascular Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ir-CPI (Experimental): Ir-CPI will be administered on top of standard of care
  Interventions: Drug: Ir-CPI
- Standard care (No Intervention): Only standard of care

INTERVENTIONS:
Drug: Ir-CPI — Participants receive a single intravenous dose of Ir-CPI during 48 hours
  Arms: Ir-CPI

SUMMARY:
The purpose of the study is to provide a first assessment of safety, tolerability and efficacy of Ir-CPI, administered on top of standard-of-care, on secondary brain injury in patients with spontaneous intracerebral haemorrhage.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients aged ≥ 18 years.
* Written informed consent obtained before any study assessment. If the patient is not able to give the informed consent personally, consent by a legal representative as defined by local law and regulation is acceptable.
* First-ever, spontaneous, supratentorial intracerebral haemorrhage in cerebral cortex or deep brain structures (putamen, thalamus, caudate, and associated deep white matter tracts) with a volume ≥ 5 mL and ≤ 60 mL determined by non-contrast CT scan.
* Patients with Glasgow Coma Scale (GCS) best motor score no less than 5.
* Modified Rankin Scale (mRS) score 0-2 prior to ICH symptom onset.

Exclusion Criteria:

* History of personal or familial bleeding disorders; including prolonged or unusual bleeding.
* Known deficiency in factor XII (FXII) or haemophilia type A (FVII) or type B (FIX) or type C (FXI).
* Infratentorial (midbrain, pons, medulla, or cerebellum) ICH.
* Secondary ICH due to aneurysm, brain tumour, arteriovenous malformation, thrombocytopenia, coagulopathy, acute sepsis, traumatic brain injury (TBI), or disseminated intravascular coagulation (DIC).
* Planned neurosurgical hematoma evacuation or other urgent surgical intervention (i.e., surgical relief of increased intracranial pressure) on initial presentation.
* Anticoagulation reversal treatment.
* Patients with intraventricular haemorrhage (IVH) having a Graeb score of >3 on initial presentation. Patients must not have blood in the 4th ventricle and may only have blood in the 3rd ventricle in the absence of ventricular expansion. Trace or mild haemorrhage in either or both lateral ventricles is permitted. Patients with hydrocephalus determined radiologically on initial presentation are excluded regardless of Graeb score.
* Use of immunosuppressive or immune-modulating therapy at admission (e.g., steroids, methotrexate, monoclonal antibodies, etc).
* Patients with active systemic bacterial, viral or fungal infections.
* Women of childbearing potential.
* Have a body weight > 120 kg at screening.
* Severe renal impairment (eGFR < 30 mL/min/1.73 m2).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2023-11-17 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events | 360 days post-randomization
Incidence of abnormalities in physical examination | 7 days post-randomization
  A complete physical examination will include, at a minimum, assessments of the cardiovascular, respiratory, gastrointestinal, dermatological, neurological (including basic neurological testing for isocoria, light reflexes, gait and balance), musculoskeletal and lymphatic systems, in addition to head, eyes, ears, nose, throat, and neck.
Change from baseline in HR interval | 7 days post-randomization
  Measured by standard 12-lead ECG
Change from baseline in PR interval | 7 days post-randomization
  Measured by standard 12-lead ECG
Change from baseline in QRS duration | 7 days post-randomization
  Measured by standard 12-lead ECG
Change from baseline in QRS axis | 7 days post-randomization
  Measured by standard 12-lead ECG
Change from baseline in QT interval | 7 days post-randomization
  Measured by standard 12-lead ECG. Two corrections of the QT interval will be investigated: Fridericia's correction (QTcF) and Bazett's correction (QTcB)
Change from baseline in blood pressure | 7 days post-randomization
  Blood pressure (systolic and diastolic) is measured using an automatic device
Change from baseline in heart rate | 7 days post-randomization
  Heart rate is measured using an automatic device
Change from baseline in body temperature | 7 days post-randomization
  Measurement of tympanic temperature

SECONDARY OUTCOMES:
Change from baseline in perihematomal oedema (PHO) and haemorrhage volumes | 10 days post-randomization
  CT scans will be acquired by volumetric CT acquisition with reconstructions in 3 planes, in order to assess hematoma volume and perihematomal volume. Assessment of hematoma expansion will be performed by comparing follow-up CT scans with baseline CT.
Measurement of the effect of Ir-CPI on the activated Partial Thromboplastin Time (aPTT) | 7 days post-randomization
  Activated partial thromboplastin time (aPTT) will be used as a pharmacodynamic marker
Measurement of the effect of Ir-CPI on the inhibition of Factor XI (FXI) and Factor XII (FXII) procoagulant activities | 7 days post-randomization
  The inhibition of Factor XI (FXI) and Factor XII (FXII) procoagulant activities will be assessed to support the aPTT dynamics
Change from baseline in Ir-CPI plasma concentrations | 7 days post-randomization

CONTACTS AND LOCATIONS:
Locations (10):
- Belgium (10):
  - HUB Erasme, Brussels, Brussels Capital
  - UCL St Luc, Brussels, Brussels Capital
  - UZ Brussel, Brussels, Brussels Capital
  - UZ Gent, Ghent, East Flanders
  - UZ Leuven, Leuven, Flemish Brabant
  - CHU Ambroise Paré, Mons, Hainaut
  - AZ Sint-Jan, Bruges, West Flanders
  - AZ Groeninge, Kortrijk, West Flanders
  - AZ Damiaan, Ostend, West Flanders
  - Clinique CHC MontLégia, Liège

IPD SHARING:
Plan to Share IPD: No